CLINICAL TRIAL: NCT04322097
Title: Characterizing Mechanisms of Upper Airway Obstruction During Drug-Induced Sleep Endoscopy (DISE)
Brief Title: Mechanisms of Upper Airway Obstruction
Acronym: DISE-CAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Raj Dedhia, MD, Associate Professor, Director, Division of Sleep Surgery, University of Pennsylvania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 833511
Record Dates: First submitted 2020-03-19; First posted 2020-03-26 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: upper airway; pharynx; collapsibility; compliance; drug-induced sleep endoscopy; hypoglossal stimulation
MeSH Terms: conditions — Sleep Apnea, Obstructive; Patient Compliance

STUDY DESIGN:
Masking Description: Participants and investigators are aware of intervention status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Study A - Functional Phenotyping during DISE (No Intervention): Participants with diagnosed OSA undergo Drug-Induced Sleep Endoscopy (DISE) to characterize determinants of upper airway obstruction using CPAP and pharyngeal manometry. Jaw thrust and other positional maneuvers are performed during DISE as part of routine clinical standard of care.
- Study B - HGNS Responders (Experimental): Participants with implanted Inspire HGNS devices undergo DISE and overnight polysomnography to assess upper airway responses with and without HGNS stimulation. CPAP titration is performed during DISE. Upper airway MRI and tongue force assessments are also conducted. Response was defined by a ≥ 50% reduction in AHI with stimulation.
  Interventions: Device: Hypoglossal Nerve Stimulation
- Study B - HGNS Nonresponders (Experimental): Participants with implanted Inspire HGNS devices undergo DISE and overnight polysomnography to assess upper airway responses with and without HGNS stimulation. CPAP titration is performed during DISE. Upper airway MRI and tongue force assessments are also conducted. Nonresponse was defined by a < 50% reduction in AHI with stimulation.
  Interventions: Device: Hypoglossal Nerve Stimulation

INTERVENTIONS:
Device: Hypoglossal Nerve Stimulation — On/off responses will be assessed both during Drug-Induced Sleep Endoscopy (DISE) and Polysomnography (PSG).
  Arms: Study B - HGNS Nonresponders; Study B - HGNS Responders

SUMMARY:
The current study is designed to examine underlying mechanisms of action of lingual muscles in the maintenance of airway patency during sleep. The investigators' major hypothesis is that specific tongue muscles are responsible for relieving upper airway obstruction during sleep.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is characterized by recurrent upper airway obstruction due to inadequate muscle tone during sleep leading to nocturnal hypercapnia, repeated oxyhemoglobin desaturations and arousals. Continuous positive airway pressure (CPAP) is the therapeutic mainstay for OSA, but adherence remains poor. The loss of motor input to the tongue during sleep has been implicated as a cause for upper airway collapse. Activation of tongue muscles with implanted hypoglossal nerve stimulators is an effective therapy for some OSA patients. Nevertheless, approximately 1/3 of OSA patients did not respond to hypoglossal nerve stimulation despite rigorous selection criteria, leaving large segments of CPAP intolerant patients at risk for OSA-related morbidity. Thus, there is a critical knowledge gap in the role of lingual muscle activity in the maintenance of airway patency.

The current study is designed to examine underlying mechanisms of action of lingual muscles in the maintenance of airway patency during sleep. The investigators' major hypothesis is that specific tongue muscles are responsible for relieving upper airway obstruction during sleep. To address this hypothesis, the investigators will (1) selectively stimulate specific lingual muscle groups (viz., protrudors and retractors) and measure effects on airway patency during Drug Induced Sleep Endoscopy (DISE). The investigators will (2) correlate responses in patency to alterations in tongue morphology (as assessed with ultrasound imaging). The investigators will (3) examine the impact of anatomic factors (e.g., the size of the maxillo-mandibular enclosure) on airway responses to stimulation. Patients will (4) undergo magnetic resonance imaging (MRI) determine the extent to which maxillo-mandibular size and tongue size and fat content compress pharyngeal structures. The investigators will (5) assess apnea severity and hypoglossal nerve stimulation with Inspire to measure response to therapy via split-night PSGs. The investigators will (6) examine digital morphometrics to quantify pharyngeal anatomy. A final goal is to (7) measure tongue force, as tongue force measurements may elucidate mechanisms of therapy response as related to neuromuscular control.

The study will contain two distinct pathways, Study A and Study B, in order to efficiently execute the protocol. Study A will focus primarily on measurements obtained as part of routine clinical care. Study B will focus on enhanced imaging and physiology techniques in patients using lingual muscle stimulation (Inspire).

Study A:

* To determine the contribution of defects in upper airway function to the pathogenesis of airway obstruction at specific sites of pharyngeal collapse by characterizing upper airway pressure-flow/area relationships during DISE.
* To determine the impact of jaw thrust and mouth closure maneuvers to functional determinants of upper airway obstruction at specific sites of pharyngeal collapse.
* To examine effects of maxillo-mandibular restriction and tongue size on upper airway functional properties during DISE.

Study B (In addition to the objectives for Study A):

* To assess effects of stimulating specific lingual muscles on upper airway patency during natural sleep and drug-induced sleep
* To assess whether craniofacial morphology predicts improvements in pharyngeal patency during sleep with stimulation.

ELIGIBILITY:
Study A Inclusion Criteria:

• Scheduled to undergo DISE as part of routine clinical standard of care.

Study B Inclusion Criteria:

* Adults (≥ 22yrs) willing and capable of providing informed consent
* Implanted with the MRI-conditional Inspire hypoglossal nerve stimulator (Model 3028 or later)
* Compliant with Inspire therapy (> 20 hours/week over 2+ weeks) as a standalone treatment for sleep-disordered breathing
* Inspire remote model 2500 or later.

Study B Exclusion Criteria:

* MRI contraindications (claustrophobia, ferromagnetic implants/foreign bodies, etc.)
* Inspire Implant Model 3024
* Inspire Remote Model 3032
* Patients who have fallen asleep while during resulting in an accident or "near miss" accident within 1 year prior to device implantation.
* Inability to sleep in the supine position (by self-report)
* History of severe difficulty initiating or maintaining sleep in the laboratory
* Pregnant women

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raj C Dedhia, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Pennsylvania Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Information from the lingual muscle stimulation arm was shared with the National Sleep Research Resource.
Time Frame: As of July, 2025, all data has been transmitted to NSRR.
Access Criteria: See criteria at the URL below.
URL: https://sleepdata.org/datasets/disecad/pages/README.md

RESULTS

PARTICIPANT FLOW:
Groups:
- Study B - Hypoglossal Nerve Stimulation (HGNS) Patients: Participants with implanted Inspire HGNS devices undergo DISE and overnight polysomnography to assess upper airway responses with and without HGNS stimulation. CPAP titration is performed during DISE. Upper airway MRI imaging and tongue force assessments are also conducted.
Period: Overall Study
Arm/Group | Study A - Functional Phenotyping During DISE | Study B - Hypoglossal Nerve Stimulation (HGNS) Patients
Started | 100 | 33
Completed | 100 | 32
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Study B - HGNS Responders: Therapy response is defined as a ≥ 50% reduction in baseline AHI with HGNS, measured during overnight polysomnography.
- Study B - HGNS Nonresponders: Therapy response is defined as a < 50% reduction in baseline AHI with HGNS, measured during overnight polysomnography.
- Total: Total of all reporting groups
Arm/Group | Study A - Functional Phenotyping During DISE | Study B - HGNS Responders | Study B - HGNS Nonresponders | Total
Number analyzed (Participants) | 100 | 13 | 19 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (14.3) | 62.4 (10.5) | 66.2 (7.2) | 57.2 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 10 | 9 | 42
  Male | 77 | 3 | 10 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 94 | 13 | 18 | 125
  Unknown or Not Reported | 5 | 0 | 0 | 5
Apnea-Hypopnea Index (AHI) [Mean (Standard Deviation); unit: events/hr] — An event is categorized as a cessation in breathing for greater than or equal to 10 seconds. AHI is calculated as a sum of all sleep-related disordered breathing events, divided by total sleep time (events/hr). Population: Three participants in study A did not have baseline sleep studies available for review.
  events/hr
    number analyzed (Participants) | 97 | 13 | 19 | 129
    (all) | 31.2 (21.1) | 37.5 (30.0) | 40.1 (19.5) | 33.2 (22.0)
BMI [Mean (Standard Deviation); unit: kg/m^2] — kg/m^2 Population: One participant in study A did not have BMI data collected.
  kg/m^2
    number analyzed (Participants) | 99 | 13 | 19 | 131
    (all) | 29.6 (4.8) | 26.6 (3.0) | 29.3 (3.7) | 29.3 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Pharyngeal Critical Pressure (Pcrit)
Description: Upper airway collapsibility (Pcrit, cmH₂O): Pressure at which the upper airway closes during inspiration, with a higher value indicating greater collapsibility.
  Pcrit less than zero indicates that the airway remains open. Pcrit greater than or equal to zero indicates that the airway is closed.
Time Frame: Collected during drug-induced sleep endoscopy (<1 day).
Population: Pcrit was unable to be measured in 20 patients (study A) and 2 patients (study B) due to technical issues and protocol deviations.
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Study A - Functional Phenotyping During DISE | Study B - HGNS Responders | Study B - HGNS Nonresponders
Number analyzed (Participants) | 80 | 12 | 18
cm H2O | 1.26 (3.29) | -1.42 (4.36) | -1.06 (2.62)
Statistical Analysis 1: Comparison: Study B - HGNS Responders vs Study B - HGNS Nonresponders; Test type: Equivalence — Alpha = 0.05; p = .80, t-test, 2 sided

2. Primary Outcome: Pharyngeal Opening Pressure (PhOP)
Description: Measurement of upper airway collapsibility (cmH2O)
Time Frame: Collected during drug-induced sleep endoscopy (<1 day).
Population: PhOP could not be obtained in 16 subjects (14 in study A, 2 for study B) due to technical issues or protocol deviations.
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Study A - Functional Phenotyping During DISE | Study B - HGNS Responders | Study B - HGNS Nonresponders
Number analyzed (Participants) | 86 | 12 | 18
cm H2O | 7.99 (3.45) | 7.33 (3.60) | 7.44 (4.08)
Statistical Analysis 1: Comparison: Study B - HGNS Responders vs Study B - HGNS Nonresponders; Test type: Equivalence — Alpha = 0.05; p = 0.94, t-test, 2 sided

3. Primary Outcome: Pharyngeal Compliance
Description: Pressure-area relationships
Time Frame: Unable to be determined
Population: Pharyngeal compliance was not analyzed from any participant due to the inability to reliably identify and standardize airway dimensions following data acquisition. Although data acquisition was performed, measurement values were not collected. Calibration was unsuccessful, and the variability in anatomical landmarks prevented a reproducible method. No valid outcome data were generated. There are no plans to further validate the measurement procedure or to analyze these data in the future.
Groups:
- Study B - HGNS Responders: Hypoglossal Nerve Stimulation: On/off responses will be assessed both during Drug-Induced Sleep Endoscopy (DISE) and Polysomnography (PSG). Response was defined by a ≥ 50% reduction in AHI with stimulation.
- Study B - HGNS Nonresponders: Hypoglossal Nerve Stimulation: On/off responses will be assessed both during Drug-Induced Sleep Endoscopy (DISE) and Polysomnography (PSG). Nonresponse was defined by a < 50% reduction in AHI with stimulation.
Arm/Group | Study A - Functional Phenotyping During DISE | Study B - HGNS Responders | Study B - HGNS Nonresponders
Number analyzed (Participants) | 0 | 0 | 0

4. Other Pre Specified Outcome: Tongue Force - Maximum
Description: Tongue force was measured using the Iowa Oral Performance Instrument (IOPI) by recording the maximum pressure generated during a 2-second sustained tongue press against a bulb. Three trials were conducted and the average value was reported for all successful trials.
Time Frame: Assessed at a single visit
Population: Tongue force was only conducted during study B.
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Study A - Functional Phenotyping During DISE | Study B - HGNS Responders | Study B - HGNS Nonresponders
Number analyzed (Participants) | 0 | 10 | 12
kPa |  | 38.0 (18.8) | 47.4 (10.9)

5. Other Pre Specified Outcome: Tongue Force - Fatigue
Description: Tongue fatigue was assessed by having participants apply maximum force to a pressure transducer and attempting to maintain this for 35 seconds. Data for each participant were reported as the time it takes for force to reduce by 67% of the maximum tongue force during each individual trial. Fatigue was reported as an average across up to 3 technically valid trials.
  Fatigue was determined by fitting a single term exponential curve to the pressure data starting at the maximal pressure (start period) and the pressure at the end of the trial.
Time Frame: Assessed at a single visit
Population: Tongue fatigue was assessed during study B only.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Study A - Functional Phenotyping During DISE | Study B - HGNS Responders | Study B - HGNS Nonresponders
Number analyzed (Participants) | 0 | 10 | 13
seconds |  | 11.1 (9.5) | 17.1 (12.7)

6. Post Hoc Outcome: Soft Palate Volume
Description: Soft palate volume measured via MRI.
Time Frame: Assessed at a single visit
Population: MRI was performed on participants in study B only, per protocol.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Study A - Functional Phenotyping During DISE | Study B - HGNS Responders | Study B - HGNS Nonresponders
Number analyzed (Participants) | 0 | 13 | 18
mm^3 |  | 9011.37 (1904.12) | 11094.10 (2721.72)

7. Post Hoc Outcome: Tongue Volume
Description: Tongue volume measured via MRI
Time Frame: Assessed at a single visit
Population: MRI was performed on participants in study B only, per protocol.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Study A - Functional Phenotyping During DISE | Study B - HGNS Responders | Study B - HGNS Nonresponders
Number analyzed (Participants) | 0 | 13 | 18
mm^3 |  | 85131.9 (16334.92) | 85322.08 (12149.09)

ADVERSE EVENTS:
Time Frame: Data were collected over the course of active participation in the trial which lasted on average 7-14 days.
Description: Adverse events were monitored through routine clinical care rather than a study-specific systematic assessment. Only events actively collected as adverse events were eligible for ClinicalTrials.gov reporting. Mild expected propofol effects and discomfort observed in routine care were not collected as adverse events and therefore were not included. No serious adverse events or deaths occurred.
Groups:
- Study B - Hypoglossal Nerve Stimulation (HGNS) Patients: Participants with implanted Inspire HGNS devices undergo DISE and overnight polysomnography to assess upper airway responses with and without HGNS stimulation. CPAP titration is performed during DISE. Upper airway MRI and tongue force assessments are also conducted.
  Hypoglossal Nerve Stimulation: On/off responses will be assessed both during Drug-Induced Sleep Endoscopy (DISE) and Polysomnography (PSG).
Arm/Group | Study A - Functional Phenotyping During DISE | Study B - Hypoglossal Nerve Stimulation (HGNS) Patients
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/32
Other Adverse Events (participants affected / at risk) | 0/100 | 0/32

LIMITATIONS AND CAVEATS:
Recruitment for Study B was delayed by COVID-19, impacting sample size and timelines.

Technical difficulties prevented pressure-area measurements in all participants.

Digital morphometrics were uninterpretable; detailed MRI scans provided a more accurate assessment of craniofacial and tongue anatomy.

Data are presented as mean (SD) with t-tests (stratified by responder status), as limited sample size restricted adherence to the original statistical plan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT04322097/Prot_001.pdf
  • Statistical Analysis Plan (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT04322097/SAP_002.pdf